CLINICAL TRIAL: NCT00300508
Title: A Randomized, Open, Comparative Multicentre Trial of 3 Years Anastrozole Treatment vs. 3 Years no Treatment in Postmenopausal Patients With Breast Cancer Who Have Completed 5 Years Adjuvant Hormone Therapy.
Brief Title: 3 Years of Anastrozole vs. no Treatment as Extended Adjuvant Therapy for Postmenopausal Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1033AU/0001; ABCSG 6A
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Breast Neoplasms
Keywords: Hormone receptor positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

INTERVENTIONS:
Drug: Anastrozole

SUMMARY:
The study assesses the effect of a further 3 years adjuvant treatment with anastrozole vs. an untreated control group after initial 5 years of adjuvant hormone-therapy.

ELIGIBILITY:
Inclusion Criteria:

* No disease recurrence at time of randomization,
* patients with breast cancer after surgery,
* 5 years (+/- 12 months) of prior endocrine therapy

Exclusion Criteria:

* Premenopausal patients,
* unknown or negative receptor status,
* Secondary malignant tumor

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 856
Dates: Start 1996-01

PRIMARY OUTCOMES:
Recurrence-free and overall survival

SECONDARY OUTCOMES:
Secondary cancers

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Austria Medical Director, MD, Study Director — AstraZeneca
Locations (51):
- Austria (51):
  - Research Site, Amstetten
  - Research Site, Bad Ischl
  - Research Site, Baden
  - Research Site, Bregenz
  - Research Site, Bruck an der Mur
  - Research Site, Dornbirn
  - Research Site, Eisenstadt
  - Research Site, Feldbach
  - Research Site, Feldkirch
  - Research Site, Freistadt
  - Research Site, Fürstenfeld
  - Research Site, Graz
  - Research Site, Güssing
  - Research Site, Hainburg an der Donau
  - Research Site, Hartberg
  - Research site, Hollabrunn
  - Research Site, Horn
  - Research Site, Innsbruck
  - Research Site, Kirchdorf
  - Research Site, Klagenfurt
  - Research Site, Klosterneuburg
  - Research Site, Krems
  - Research Site, Kufstein
  - Research Site, Leoben
  - Research Site, Linz
  - Research Site, Mistelbach
  - Research Site, Mödling
  - Research Site, Neunkirche
  - Research Site, Oberpullendorf
  - Research Site, Oberwart
  - Research Site, Ried im Innkreis
  - Research Site, Rohrbach
  - Research Site, Rottenmann
  - Research Site, Salzburg
  - Research Site, Sankt Pölten
  - Research Site, Sankt Veit an der Glan
  - Research Site, Schärding
  - Research Site, Scheibbs
  - Research Site, Schladming
  - Research Site, Schwarzach
  - Research Site, Spittal an der Drau
  - Research Site, Steyr
  - Research Site, Tulln
  - Research Site, Vienna
  - Research Site, Villach
  - Research Site, Vöcklabruck
  - Research Site, Waidhofen an der Ybbs
  - Research Site, Wels
  - Research Site, Wiener Neustadt
  - Research Site, Wolfsberg
  - Research Site, Zams

REFERENCES:
- [Derived] Wimmer K, Hlauschek D, Balic M, Pfeiler G, Greil R, Singer CF, Halper S, Steger G, Suppan C, Gampenrieder SP, Helfgott R, Egle D, Filipits M, Jakesz R, Solkner L, Fesl C, Gnant M, Fitzal F. Is the CTS5 a helpful decision-making tool in the extended adjuvant therapy setting? Breast Cancer Res Treat. 2024 Jun;205(2):227-239. doi: 10.1007/s10549-023-07186-6. Epub 2024 Jan 25. PMID 38273214
- [Derived] Gnant M, Pfeiler G, Stoger H, Mlineritsch B, Fitzal F, Balic M, Kwasny W, Seifert M, Stierer M, Dubsky P, Greil R, Steger G, Samonigg H, Fesl C, Jakesz R. The predictive impact of body mass index on the efficacy of extended adjuvant endocrine treatment with anastrozole in postmenopausal patients with breast cancer: an analysis of the randomised ABCSG-6a trial. Br J Cancer. 2013 Aug 6;109(3):589-96. doi: 10.1038/bjc.2013.367. Epub 2013 Jul 18. PMID 23868011